CLINICAL TRIAL: NCT05788809
Title: Communication Skill and Related Factors Among Oncology Nurses
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202301188RIND; 23MMHIS49e (Other: Mackay Memorial Hospital Institutional Review Board)
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2023-08

CONDITIONS: Oncology; Nurse; Communication
Keywords: Oncology nurse; Communication skill
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a 1-year quantitative method research.Data collection will be divided into oncology nurses and cancer patients.To explore the related factors of clinical oncology nurses on the psychological aspects of cancer patients.

DETAILED DESCRIPTION:
Background:Nurses who care for cancer patients on the front line play an important role in the psychological care, distress assessment and management of cancer patients. Most of these cancer patients do not directly express their concerns to the nursing staff. Nursing staff should be able to assess and identify psychological needs through verbal and non-verbal messages during the nursing period, and provide effective information, general psychological support and rich psychological support in nursing measures. The ability to communicate empathetically and avoid ignoring psychological needs that may cause distress to the patient. Therefore, an in-depth understanding of the first-line tumor nurses interacting with patients, and the related factors that affect communication with patients, such as workload, fatigue, self-confidence, etc., are crucial factors for detecting psychological problems in cancer patients. It directly affects the body and mind of cancer patients, and exploring its related factors is of course an important topic.

Purpose: Understand current clinical oncology nurses, work load, emotional state, self-confidence, comfort ability, empathy and communication ability related factors, and add patients' measurement of nursing staff's communication ability, empathy and satisfaction, through nurses The results of the patients and nurses are closer to the current clinical situation.

Method:This study is a 1-year quantitative method research. It is a cross-sectional descriptive correlation research, using a structured questionnaire to collect data which will be collected by oncology nurses and cancer patients.

ELIGIBILITY:
Nurse

Inclusion Criteria:

* Over 20 years old (inclusive).
* Nursing staff who are currently working in cancer-related positions and have clinical contact or care for patients.

Exclusion Criteria:

* Nurse who have resigned.

Patient

Inclusion Criteria:

* Over 20 years old (inclusive).
* Diagnosed as a cancer patient by doctors.
* Patients who are known disease status.
* Patients who are currently hospitalized in cancer wards.

Exclusion Criteria:

* People with mental illness.
* Those who are unconscious and unable to complete the interview for this study with language or conversation.
* Those who are unwilling to accept interviews and participate in research surveys.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurse who are over 20 years old (inclusive) and care cancer patients currently. Patient who are over 20 years old (inclusive) and diagnosed with cancer.
Sampling Method: Non-Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Communication skills | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Oncology nurses' communication skills were measured by Communication Skills in Health Professionals (CSS-HP) in nurse's questionnaire which is a 6 Liker scale(1-6). Also,communication skills were measured by Communication Assessment Tool (CAT) in patient's questionnaire which is a 5 Liker scale(1-5). Both of scales are higher scores representing better communication skills.

SECONDARY OUTCOMES:
Physical and Psychological state scale | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Oncology nurse's physical and psychological state will be measured by NRS(0-10). Item contains work loading,burn out feeling and degree of distress.The higher the score, the more work loading,burn out feeling or degree of distress you have.
The pressure source of work | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Oncology nurse's pressure source will be measured by Work Stressor Inventory for Nurses in Oncology (WSINO) which is a 5-Point Likert Scale(1-5). The higher the score, the more frequently the question occurs.
Self efficacy scale (GSES) | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Oncology nurses' self-efficacy were measured by self efficacy scale. It's a 4 point (1-4),higher the score means the more confident you have. There is also 11 point (0-10) scale that higher the score means the more confident you are in caring for patients.
Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being (FACIT-Sp) | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Oncology nurses' spiritual well-being were measured by FACIT-Sp.It is a 5 Liker scale(0-4),higher scores represent better well-being.
Efferson Empathy Scale | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Oncology nurses' empathy will be measured by Efferson Empathy Scale in nurse's questionnaire. It is a 7 Liker scale(1-7),higher scores means someone have more empathy on caring patients.Also,in patient's questionnaire that nurses' empathy were measured by Self-created questionnaire which is a 7 Liker scale(1-7),higher scores mean patients feel more empathy.
Newcastle Satisfaction with Nursing Scale(NSNS) | 1 time points: From date of approaching patient until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Patient satisfaction with nursing care will be measured by NSNS.It is a 5 Liker scale(1-5),higher scores mean patients feel more satisfaction .

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan